CLINICAL TRIAL: NCT01923181
Title: Multiple Dose Trial Examining Dose Range, Escalation and Efficacy of Oral Semaglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-3790; 2012-004994-16 (EudraCT Number); U1111-1136-4716 (Other: WHO)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1:Semaglutide tablets : 2.5 mg (Experimental): 2.5 mg for 26 weeks. All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 2:Semaglutide tablets: 2.5 mg/5 mg (Experimental): 2.5 mg for 4 weeks, then 5.0 mg for 22 weeks. All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 3:Semaglutide tablets: 5.0 mg/10 mg (Experimental): 5.0 mg for 4 weeks, then 10 mg for 22 weeks. All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 4:Semaglutide tablets:5.0 mg/10 mg/20 mg (Experimental): 5.0 mg for 4 weeks, then 10 mg for 4 weeks, then 20 mg for 18 weeks. All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 5:Semaglutide tablets:5.0 mg/10 mg/20 mg/40 mg (Experimental): 5.0 mg for 4 weeks, then 10 mg for 4 weeks, then 20 mg for 4 weeks, then 40 mg for 14 weeks.
  All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 6:Semaglutide tablets:5.0 mg/10 mg/20 mg/40 mg (Experimental): 5.0 mg for 8 weeks, then 10 mg for 8 weeks, then 20 mg for 8 weeks, then 40 mg for 2 weeks All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 7:Semaglutide tablets: 5.0 mg/10 mg/20 mg/40 mg (Experimental): 5.0 mg for 2 weeks, then 10 mg for 2 weeks, then 20 mg for 2 weeks, then 40 mg for 20 weeks.
  All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide
- 8:Placebo tablets (Placebo Comparator): All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: oral placebo
- 9:Semaglutide injections :0.25 mg/0.50 mg/1.0 mg (Active Comparator): 0.25 mg for 4 weeks, then 0.50 mg for 4 weeks, then 1.0 mg for 18 weeks. All arms include 26 weeks of treatment and a 5 week follow-up period. The trial medication will be add-on to metformin therapy or as monotherapy in the case where the subject is treated with diet and exercise alone.
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Once-daily oral administration as tablets.
  Arms: 1:Semaglutide tablets : 2.5 mg; 2:Semaglutide tablets: 2.5 mg/5 mg; 3:Semaglutide tablets: 5.0 mg/10 mg; 4:Semaglutide tablets:5.0 mg/10 mg/20 mg; 5:Semaglutide tablets:5.0 mg/10 mg/20 mg/40 mg; 6:Semaglutide tablets:5.0 mg/10 mg/20 mg/40 mg; 7:Semaglutide tablets: 5.0 mg/10 mg/20 mg/40 mg
Drug: semaglutide — Once-weekly,injected s.c./subcutaneously (under the skin) using a pen
  Arms: 9:Semaglutide injections :0.25 mg/0.50 mg/1.0 mg
Drug: oral placebo — Once-daily oral administration as tablets.
  Arms: 8:Placebo tablets

SUMMARY:
This trial is conducted globally. The aim of the trial is to examine the dose range, escalation and efficacy of oral semaglutide in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI above or equal to 25 and below or equal to 40 kg/m^2
* Subjects diagnosed with T2D (Type 2 diabetes) treated with diet and exercise and/or who have been on a stable dose of metformin for at least 30 days prior to screening
* HbA1c 7.0-9.5% (53-80 mmol/mol) (both inclusive)

Exclusion Criteria:

* Subjects on selected oral medication with a narrow therapeutic window, such as warfarin, digoxin, tricyclic antidepressants, lithium, aminophylline, theophylline and anticonvulsants
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Chronic malabsorption, regardless of aetiology
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Treatment with glucose lowering agent(s) other than metformin as stated in the inclusion criteria in a period of 90 days before the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2014-12-11 (Actual); Study Completion 2014-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (94):
- United States (37):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, South Miami, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Addison, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Jersey Shore, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Spring Hill, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Wenatchee, Washington
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Saint Stefan
  - Novo Nordisk Investigational Site, Vienna
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Canada (6):
  - Novo Nordisk Investigational Site, Bathurst, New Brunswick
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Stayner, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
- Denmark (6):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Svendborg
- Germany (7):
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Speyer
- Israel (7):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Herzliya
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
- Italy (4):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Verona
- Malaysia (4):
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Ipoh
  - Novo Nordisk Investigational Site, Kota Bharu
  - Novo Nordisk Investigational Site, Seri Manjung
- Novo Nordisk Investigational Site, Belgrade, Serbia
- South Africa (2):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
- Spain (4):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Sweden (4):
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Oskarshamn
  - Novo Nordisk Investigational Site, Örebro
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Chesterfield, Derbyshire
  - Novo Nordisk Investigational Site, Crewe
  - Novo Nordisk Investigational Site, Hinckley
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London

REFERENCES:
- [Result] Davies M, Pieber TR, Hartoft-Nielsen ML, Hansen OKH, Jabbour S, Rosenstock J. Effect of Oral Semaglutide Compared With Placebo and Subcutaneous Semaglutide on Glycemic Control in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA. 2017 Oct 17;318(15):1460-1470. doi: 10.1001/jama.2017.14752. PMID 29049653
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 100 sites in 14 countries as follows: Austria (6), Bulgaria (3), Canada (6), Denmark (6), Germany (6), Israel (6), Italy (4), Malaysia (4), Serbia (1), South Africa (3), Spain (5), Sweden (3), United Kingdom (8) and United States (39).
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 2.5 mg: Participants were to take 2.5 mg oral semaglutide tablets once daily for 26 weeks. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 5 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 2.5 mg from week 1 to 4 and 5 mg from week 5 to 26. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 10 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 5 mg from week 1 to 4 and 10 mg from week 5 to 26. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 20 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 5 mg from week 1 to 4, 10 mg from week 5 to 8 and 20 mg from week 9 to 26.
  Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 40 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 5 mg from week 1 to 4, 10 mg from week 5 to 8, 20 mg from week 9 to 12 and 40 mg from week 13 to 26. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 40 mg Slow Dose-escalation: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 5 mg from week 1 to 8, 10 mg from week 9 to 16, 20 mg from week 17 to 24 and 40 mg from week 25 to 26. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets.
- Oral Semaglutide 40 mg Fast Dose-escalation: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 26: 5 mg from week 1 to 2, 10 mg from week 3 to 4, 20 mg from week 5 to 6 and 40 mg from week 7 to 26. Semaglutide tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than semaglutide tablets could be taken upto 2 hours prior to administration of semaglutide tablets. The semaglutide tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide tablets. Oral medication other than semaglutide tablets could only be taken 2 hours after administration of semaglutide tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide tablets
- Subcutaneous Semaglutide 1 mg: Participants were to administer subcutaneous semaglutide injections once weekly in a dose escalation manner from week 1 to 26: 0.25 mg from week 1 to 4, 0.50 mg from week 5 to 8 and 1.0 mg from week 9 to 26. Semaglutide injections were to be administered in the thigh, abdomen or upper arm, at any time of day (same day of the week) irrespective of meals.
- Placebo: Participants were to take oral semaglutide placebo tablets once daily from week 1 to 26. Semaglutide placebo tablets were to be taken once daily in the morning in a fasting state (atleast for 6 hours). Water and oral medication other than the semaglutide placebo tablets could be taken upto 2 hours prior to administration of semaglutide placebo tablets. The semaglutide placebo tablets could be taken with up to 120 mL of water. Participants were not allowed to take food and water for at least 30 minutes after administration of semaglutide placebo tablets. Oral medication other than semaglutide placebo tablets could only be taken 2 hours after administration of semaglutide placebo tablets. If taken along with food, oral medication could be administered 30 minutes after administration of semaglutide placebo tablets.
Period: Overall Study
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Started | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71
Full Analysis Set (FAS) | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71
Safety Analysis Set (SAS) | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71
Completed | 67 | 64 | 67 | 65 | 63 | 66 | 62 | 61 | 68
Not Completed | 3 | 6 | 2 | 5 | 8 | 4 | 8 | 8 | 3
Not completed — Protocol Violation | 2 | 2 | 0 | 2 | 2 | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 4 | 2 | 4 | 3 | 1
Not completed — Other | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 1 | 2 | 1 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71 | 630
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (9.9) | 55.7 (11.0) | 56.5 (10.1) | 58.3 (10.4) | 56.5 (10.2) | 57.1 (10.5) | 57.7 (10.8) | 56.8 (11.8) | 58.9 (10.3) | 57.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 26 | 26 | 28 | 29 | 26 | 21 | 31 | 235
  Male | 45 | 47 | 43 | 44 | 43 | 41 | 44 | 48 | 40 | 395
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 7 | 7 | 9 | 12 | 7 | 9 | 71
  Not Hispanic or Latino | 64 | 63 | 62 | 63 | 64 | 61 | 58 | 62 | 62 | 559
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race of participants
  Participants
    White | 57 | 63 | 57 | 59 | 63 | 54 | 59 | 54 | 57 | 523
    Black or African American | 6 | 2 | 7 | 4 | 4 | 7 | 7 | 4 | 6 | 47
    Asian | 7 | 4 | 4 | 4 | 3 | 7 | 4 | 10 | 7 | 50
    American Indian or Alaska Native | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Other | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 7
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 7.99 (0.72) | 7.80 (0.62) | 7.80 (0.70) | 7.86 (0.69) | 8.05 (0.75) | 7.96 (0.73) | 7.77 (0.75) | 7.77 (0.71) | 8.00 (0.80) | 7.89 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline (week 0) in HbA1c was evaluated at week 26. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Groups:
- Oral Semaglutide 40 mg Pooled: The data from participants in oral semaglutide 40 mg arm and oral semaglutide fast dose-escalation arm were pooled in this arm.
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Oral Semaglutide 40 mg Pooled | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 56 | 58 | 57 | 48 | 46 | 52 | 44 | 90 | 48 | 51
Percentage of HbA1c | -0.88 (0.77) | -1.23 (0.79) | -1.56 (0.92) | -1.70 (0.75) | -2.04 (0.90) | -1.76 (0.92) | -1.65 (0.77) | -1.85 (0.86) | -1.85 (0.75) | -0.40 (0.84)
Statistical Analysis 1: Comparison: Oral Semaglutide 40 mg Pooled vs Placebo; Results are based on the data from the on-treatment without rescue medication observation period. The analysis was based on mixed model for repeated measurements with treatment, stratum and country as fixed factors and baseline value as covariate, all nested within visit. Group mean estimates were adjusted according to observed baseline distribution; Test type: Superiority — This hypothesis was controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Mean treatment difference = -1.47, 95% CI 2-sided [-1.73 to -1.22] — Oral semaglutide 40 mg pooled - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 2.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0069, Mixed Models Analysis; Treatment difference = -0.40, 95% CI 2-sided [-0.69 to -0.11] — Oral semaglutide 2.5 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.89, 95% CI 2-sided [-1.18 to -0.60] — Oral semaglutide 5 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.18, 95% CI 2-sided [-1.47 to -0.90] — Oral semaglutide 10 mg - Placebo
Statistical Analysis 5: Comparison: Oral Semaglutide 20 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.38, 95% CI 2-sided [-1.68 to -1.09] — Oral Semaglutide 20 mg - Placebo
Statistical Analysis 6: Comparison: Oral Semaglutide 40 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.60, 95% CI 2-sided [-1.89 to -1.30] — Oral semaglutide 40 mg - Placebo
Statistical Analysis 7: Comparison: Oral Semaglutide 40 mg Slow Dose-escalation vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.43, 95% CI 2-sided [-1.72 to -1.14] — Oral semaglutide 40 mg slow dose-escalation - Placebo
Statistical Analysis 8: Comparison: Oral Semaglutide 40 mg Fast Dose-escalation vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.34, 95% CI 2-sided [-1.64 to -1.04] — Oral semaglutide 40 mg fast dose-escalation - Placebo
Statistical Analysis 9: Comparison: Subcutaneous Semaglutide 1 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.56, 95% CI 2-sided [-1.85 to -1.27] — Subcutaneous semaglutide 1 mg - Placebo
Statistical Analysis 10: Comparison: Oral Semaglutide 2.5 mg vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = 1.16, 95% CI 2-sided [0.87 to 1.45] — Oral semaglutide 2.5 mg - Subcutaneous semaglutide 1 mg
Statistical Analysis 11: Comparison: Oral Semaglutide 5 mg vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Mixed Models Analysis; Treatment difference = 0.67, 95% CI 2-sided [0.38 to 0.96] — Oral semaglutide 5 mg - Subcutaneous semaglutide 1 mg
Statistical Analysis 12: Comparison: Oral Semaglutide 10 mg vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0116, Mixed Models Analysis; Treatment difference = 0.37, 95% CI 2-sided [0.08 to 0.67] — Oral semaglutide 10 mg - Subcutaneous semaglutide 1 mg
Statistical Analysis 13: Comparison: Oral Semaglutide 20 mg vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.2440, Mixed Models Analysis; Treatment difference = 0.18, 95% CI 2-sided [-0.12 to 0.47] — Oral semaglutide 20 mg - Subcutaneous semaglutide 1 mg
Statistical Analysis 14: Comparison: Oral Semaglutide 40 mg vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.7973, Mixed Models Analysis; Treatment difference = -0.04, 95% CI 2-sided [-0.34 to 0.26] — Oral semaglutide 40 mg - Subcutaneous semaglutide 1 mg
Statistical Analysis 15: Comparison: Oral Semaglutide 40 mg Slow Dose-escalation vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.3901, Mixed Models Analysis; Treatment difference = 0.13, 95% CI 2-sided [-0.16 to 0.42] — Oral semaglutide 40 mg slow-dose escalation - Subcutaneous semaglutide 1 mg
Statistical Analysis 16: Comparison: Oral Semaglutide 40 mg Fast Dose-escalation vs Subcutaneous Semaglutide 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1612, Mixed Models Analysis; Treatment difference = 0.22, 95% CI 2-sided [-0.09 to 0.52] — Oral semaglutide 40 mg fast-dose escalation - Subcutaneous semaglutide 1 mg
Statistical Analysis 17: Comparison: Oral Semaglutide 40 mg vs Oral Semaglutide 40 mg Slow Dose-escalation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.2669, Mixed Models Analysis; Treatment difference = 0.17, 95% CI 2-sided [-0.13 to 0.46] — Oral semaglutide 40 mg slow-dose escalation - Oral semaglutide 40 mg
Statistical Analysis 18: Comparison: Oral Semaglutide 40 mg vs Oral Semaglutide 40 mg Fast Dose-escalation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0989, Mixed Models Analysis; Treatment difference = 0.26, 95% CI 2-sided [-0.05 to 0.56] — Oral semaglutide 40 mg fast-dose escalation - Oral semaglutide 40 mg
Statistical Analysis 19: Comparison: Oral Semaglutide 40 mg Slow Dose-escalation vs Oral Semaglutide 40 mg Fast Dose-escalation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.5565, Mixed Models Analysis; Treatment difference = 0.09, 95% CI 2-sided [-0.21 to 0.39] — Oral semaglutide 40 mg fast-dose escalation - Oral semaglutide 40 mg slow-dose escalation

2. Secondary Outcome: Subjects Who Achieve (Yes/no) HbA1c Below 7 Percent (53 mmol/Mol)
Description: Participants who achieved HbA1c <7.0%, was evaluated at week 26. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: After 26 weeks of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 56 | 58 | 57 | 48 | 46 | 52 | 44 | 48 | 51
Participants
  Yes | 27 | 50 | 49 | 41 | 42 | 47 | 38 | 45 | 18
  No | 29 | 8 | 8 | 7 | 4 | 5 | 6 | 3 | 33

3. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 47 | 46 | 51 | 44 | 46 | 51
kg | -2.01 (3.08) | -2.89 (3.32) | -4.90 (4.04) | -5.75 (5.63) | -6.91 (4.57) | -5.93 (4.34) | -8.29 (5.27) | -6.71 (3.18) | -1.16 (2.59)

4. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 26. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 56 | 56 | 57 | 47 | 46 | 51 | 44 | 46 | 51
cm | -2.00 (4.31) | -2.29 (4.54) | -5.28 (5.55) | -4.08 (4.01) | -5.71 (4.65) | -4.86 (5.48) | -6.24 (4.71) | -6.34 (4.65) | -2.29 (3.99)

5. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 26. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 47 | 46 | 51 | 44 | 46 | 51
kg/m^2 | -0.67 (0.98) | -0.98 (1.14) | -1.72 (1.44) | -1.93 (1.87) | -2.37 (1.58) | -2.04 (1.45) | -2.92 (1.93) | -2.32 (1.04) | -0.43 (0.94)

6. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Recorded
Description: TEAEs were recorded during weeks 0-31 (26 weeks treatment period+5 weeks follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all participants exposed to at least 1 dose of randomised semaglutide or placebo.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71
Events | 142 | 169 | 233 | 289 | 230 | 233 | 245 | 218 | 127

7. Secondary Outcome: Number of Confirmed Hypoglycaemic Episodes Recorded
Description: Treatment-emergent confirmed hypoglycaemic episodes were recorded during weeks 0-31 (26 weeks treatment period + 5 weeks follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Confirmed hypoglycaemic episode is an episode that is severe according to the American Diabetes Association (ADA) classification or plasma glucose value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = SAS which comprised all participants exposed to at least 1 dose of randomised semaglutide or placebo.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 70 | 70 | 69 | 70 | 71 | 70 | 70 | 69 | 71
Episodes | 4 | 4 | 6 | 1 | 1 | 3 | 1 | 6 | 5

ADVERSE EVENTS:
Time Frame: Week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 2.5 mg | Oral Semaglutide 5 mg | Oral Semaglutide 10 mg | Oral Semaglutide 20 mg | Oral Semaglutide 40 mg | Oral Semaglutide 40 mg Slow Dose-escalation | Oral Semaglutide 40 mg Fast Dose-escalation | Subcutaneous Semaglutide 1 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70 | 0/69 | 0/70 | 0/71 | 0/70 | 0/70 | 0/69 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/70 | 2/70 | 2/69 | 0/70 | 1/71 | 3/70 | 5/70 | 2/69 | 5/71
Other Adverse Events (participants affected / at risk) | 35/70 | 32/70 | 37/69 | 49/70 | 49/71 | 42/70 | 55/70 | 44/69 | 34/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 2.5 mg (N=70) | Oral Semaglutide 5 mg (N=70) | Oral Semaglutide 10 mg (N=69) | Oral Semaglutide 20 mg (N=70) | Oral Semaglutide 40 mg (N=71) | Oral Semaglutide 40 mg Slow Dose-escalation (N=70) | Oral Semaglutide 40 mg Fast Dose-escalation (N=70) | Subcutaneous Semaglutide 1 mg (N=69) | Placebo (N=71)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 2.5 mg (N=70) | Oral Semaglutide 5 mg (N=70) | Oral Semaglutide 10 mg (N=69) | Oral Semaglutide 20 mg (N=70) | Oral Semaglutide 40 mg (N=71) | Oral Semaglutide 40 mg Slow Dose-escalation (N=70) | Oral Semaglutide 40 mg Fast Dose-escalation (N=70) | Subcutaneous Semaglutide 1 mg (N=69) | Placebo (N=71)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 4 (5) | 5 (7) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 3 (3) | 3 (4) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (8) | 3 (3) | 4 (4) | 3 (3) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 6 (8) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4) | 6 (8) | 5 (8) | 9 (11) | 7 (7) | 8 (9) | 7 (7) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 10 (10) | 8 (8) | 10 (11) | 3 (4) | 11 (11) | 9 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 7 (7) | 16 (20) | 14 (18) | 10 (15) | 14 (27) | 12 (15) | 10 (14) | 7 (10)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (6) | 5 (7) | 6 (6) | 8 (8) | 6 (8) | 6 (8) | 5 (5) | 10 (11) | 3 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 3 (3) | 5 (6) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 2 (2) | 4 (6) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 5 (7) | 4 (4) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 9 (9) | 8 (10) | 10 (18) | 4 (7) | 8 (10) | 7 (7) | 10 (21) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 2 (2) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 3 (5) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (7)
Lipase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 3 (4) | 3 (3) | 5 (6) | 5 (5) | 3 (4) | 4 (5) | 2 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 9 (12) | 10 (13) | 23 (27) | 25 (37) | 24 (37) | 23 (29) | 25 (27) | 22 (23) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5) | 1 (1) | 6 (7) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8) | 4 (5) | 14 (18) | 12 (15) | 14 (25) | 11 (22) | 16 (20) | 6 (6) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT01923181/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT01923181/SAP_001.pdf